CLINICAL TRIAL: NCT00854685
Title: A Factorial-design, Randomised, Double-blind, Placebo-controlled, Dose Optimisation Study to Investigate the Safety, Efficacy, Immunogenicity and Pharmacokinetics of ART621 Following Multiple Dose Administration in Subjects Diagnosed With Rheumatoid Arthritis Concomitantly Taking Methotrexate
Brief Title: Dose Optimisation Study of ART621 in Subjects Diagnosed With Rheumatoid Arthritis Taking Methotrexate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arana Therapeutics Ltd (Industry)
Collaborators: Trident Clinical Research Pty Ltd (Industry)
Responsible Party: David Fuller, Chief Medical Officer, Arana Therapeutics Limited
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: ART621-223
Record Dates: First submitted 2009-03-01; First posted 2009-03-03 (Estimated); Last update posted 2010-01-06 (Estimated); Status verified 2009-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- 1 (Experimental)
  Interventions: Drug: ART621
- 2 (Experimental)
  Interventions: Drug: ART621
- 3 (Experimental)
  Interventions: Drug: ART621
- 4 (Experimental)
  Interventions: Drug: ART621
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo
- 6 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ART621 — 3.0mg/kg s.c. - weekly
  Arms: 1
Drug: ART621 — 3.0mg/kg s.c. - fortnightly
  Arms: 2
Drug: ART621 — 1.5mg/kg s.c. - weekly
  Arms: 3
Drug: ART621 — 1.5mg/kg s.c. - fortnightly
  Arms: 4
Drug: Placebo — Placebo s.c. - weekly
  Arms: 5
Drug: Placebo — Placebo s.c. - fortnightly
  Arms: 6

SUMMARY:
The purpose of this clinical trial is to establish what dose level and dosing frequency is optimal in the treatment of rheumatoid arthritis patients with ART621.

DETAILED DESCRIPTION:
Despite being effective in approximately 60% of subjects, there are limitations to existing anti-TNF therapies especially in relation to immunogenicity, safety and administration. In addition, due to their high molecular weight, currently marketed products are largely confined to the blood stream.

ART621 is an anti-TNF molecule that contains 2 identical domain "antibodies" that have the binding activity of a full antibody but with a substantially smaller molecular size. The molecular weight of approximately half that of full size antibodies is predicted to, a) have improved tissue penetration and, b) to be less immunogenic than full size antibodies.

This clinical trial is designed to establish the optimal dose level and dose frequency of ART621 in the treatment of patients with rheumatoid arthritis and to obtain data relating to the safety, immunogenicity and pharmacokinetics of ART621 when administered with an intravenous loading dose followed by subcutaneous administration every week compared to every fortnight.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are willing to give signed informed consent..
* Male or female subjects at least 18 years of age and no more than 80 years of age.
* Women of childbearing potential, or men of reproductive potential, must be using adequate (in the investigator's opinion) birth control measures (e.g. abstinence, oral contraceptives, intrauterine device, barrier method with spermicide, or surgical sterilisation) during the study. Female subjects of childbearing potential must test negative for pregnancy prior to enrolling in the study. Post menopausal (cessation of menses for more than 2 years) women are eligible for this study.
* Diagnosis of RA according to the revised (1987) American College of Rheumatology criteria for at least 6 months prior to screening.
* Meet ACR functional class criteria I, II or III.
* Have active RA at the time of screening and at baseline, defined as ≥ 6 swollen joints and ≥ 6 tender joints (from 68 joint count) together with at least 2 of the following 3 criteria:

  * CRP level ≥ 1.5 mg/dl;
  * ESR by Westergren method ≥ 28 mm in the first hour; or
  * morning stiffness ≥ 45 minutes.
* At least one of the following should be present at screening:

  * documented history or current presence of positive rheumatoid factor;
  * presence of serum anti-CCP antibodies; or
  * screening radiographic erosion.
* Have been tolerating concomitant methotrexate (oral or subcutaneous) for at least 3 months prior to screening and on a stable dose between 10-25 mg per week for at least 6 weeks prior to the first study dose. The route of administration must also be stable. Use of methotrexate dose of 25-50 mg every 2 weeks is also acceptable. (Other DMARDs taken concomitantly with methotrexate are not allowed. Those subjects concomitantly receiving additional DMARDs with methotrexate may enter the study by stopping the additional DMARD at least 4 weeks prior to first study dose).
* If using the following medication, the subject must be on a stable dose for the 4 weeks prior to the first study dose and maintain that dose throughout the study:

  * oral corticosteroids, equivalent to ≤ 10 mg of prednisone/day.
  * one nonsteroidal anti-inflammatory drug (NSAID).
  * 3-hydroxy-3-methylglutaryl-coenzyme A reductase inhibitors (statins) or fibrates (see Section 7.1 for acceptable doses).
* Does not have active or latent TB according to eligibility assessment and screening tests.
* Is willing and able to comply with study visits and other protocol requirements.

Exclusion Criteria:

* Body weight >98 kg.
* Pregnant, nursing, or planning a pregnancy (both men and women) within 9 months of enrolment.
* Screening laboratory tests:

  * haemoglobin ≤ 8.0 gm/dl
  * white blood cells ≤ 3.0 x103 cells/µl
  * neutrophils ≤ 1.5 x 103 cells/µl
  * platelets ≤100 x 103 cells/µl
  * serum transaminase level (AST and ALT) ≥ 2 times upper limit of normal (ULN)
  * serum creatinine ≥ 0.15 mmol/l
* Subjects with a diagnosis of juvenile arthritis or other inflammatory or autoimmune diseases that might confound the evaluations of benefit from ART621 such as ankylosing spondylitis, systemic lupus erythematosus and Lyme disease.
* Subjects who have previously failed to respond to any oral or injectable anti-TNFα therapy or subjects who have had to stop anti-TNFα therapy for safety reasons. Subjects who have successfully responded to anti-TNF therapy in the past (but discontinued for reasons other than safety or lack of efficacy) > 6 months prior to study day one may enrol. Patients who have participated in a previous anti-TNF therapy study are eligible if they are confirmed to have received placebo.
* Subjects who have previously received the following anti-rheumatic drugs: interleukin-1 receptor antagonist [anakinra], rituximab, anti-CD4 antibody, abatacept, thalidomide, p38 MAP kinase inhibitor and other agents (other than those listed in Section 7.3).
* Subjects who have undergone plasmapheresis within 6 months prior to randomisation.
* Have received intraarticular, intramuscular, or intravenous corticosteroids, including intramuscular adrenocorticotropic hormone, during the 4 weeks prior to the first study dose, or non-stable doses of oral steroids.
* Subjects with a history of any clinically significant adverse reaction to murine or chimeric proteins, including serious allergic reactions.
* Subjects with Felty's syndrome or a history of Felty's syndrome.
* Subjects who have received or are expecting to receive any live virus or bacterial vaccinations within 1 month before first study dose, during the study, or up to 3 months after the study dose.
* Subjects with a history of, presence of, or at high risk of serious infection including:

  * history of active TB, or positive Mantoux test or QuantiFERON Gold test or chest x-ray suggestive of active or healed TB or positive contact history with a subject with active TB within the past 3 months. If patients have a positive Mantoux test but a negative QuantiFERON Gold test, they may be enrolled.
  * a serious infection during the 3 months prior study entry (hospitalised or received IV antibiotics for an infection).
  * chronic or recurrent infectious disease.
  * systemic fungal infections
  * opportunistic infection within 3 months prior to screening (refer to 1993 CDC Classification System for HIV Infection).
  * subjects known, or suspected, to be infected with HIV, hepatitis B, or hepatitis C.
  * subjects with planned joint replacement surgery or a history of infected joint prosthesis or who have received antibiotics for a suspected infection of a joint prosthesis if that prosthesis has not been removed or replaced.
* Subjects with a known history of demyelinating diseases such as multiple sclerosis or optic neuritis.
* Subjects with evidence of severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic, psychiatric, or cerebral disease.
* Concurrent CHF, including medically controlled, asymptomatic CHF or ECG findings suggestive of CHF.
* Subjects receiving cytotoxic drugs including cyclophosphamide, cyclosporine, or alkylating agents within 6 months prior to first study dose.
* Known history or evidence of malignancy, lymphoproliferative or neoplastic disease with the exception of successfully treated basal or squamous cell carcinoma of the skin or cervical intraepithelial neoplasia.
* Subjects who have undergone organ transplant (with exception of a corneal transplant more than 3 months prior to screening).
* Subjects previously enrolled in this study, currently participating in another investigational study or treated with any investigational drug within the previous 3 months or within 5 half-lives, whichever is greater, prior to first study dose.
* Any other clinically significant disease or disorder or factors such as substance abuse which in the opinion of the investigator make the subject ineligible for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-02; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of subcutaneous injections of ART621 (preceded by a single i.v. loading dose) at different dose frequencies | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Rheumatology, National Hospital Sri Lanka, Colombo, Sri Lanka